CLINICAL TRIAL: NCT00522704
Title: Correlation Between Access Blood Flow and Extracorporeal Blood Flow
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Collaborators: JOSE CARRASCO ARTEAGA HOSPITAL FROM Ecuadorian Institute of Social Security (Unknown)
Responsible Party: Principal Investigator, FRANKLIN MORA, Doctor, Instituto Nacional de Cardiologia Ignacio Chavez
Other Study IDs: INCich-07-08-7403
Record Dates: First submitted 2007-08-28; First posted 2007-08-30 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Arteriovenous Fistula
Keywords: Arteriovenous fistula; Access blood flow; Extracorporeal blood flow; Dynamic arterial line pressure; Hemodialysis treatment
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Dynamic Arterial line Pressure (DALP) — eEBF will be record with dynamic arterial line pressure of -60 mmHg (eEBF-60 mmHg), -100 mmHg (eEBF-100 mmHg), -160 mmHg (eEBF-160 mmHg), -200 mmHg (eEBF-200 mmHg) and -260 mmHg (eEBF-260 mmHg) during the first one half hour of the dialysis session. Access Blood flow will be performed with blood thermal monitor.
  Other Names: BTM,

SUMMARY:
The purpose of this study is to determine if Effective Extracorporeal Blood Flow(eEBF) has correlation with Access Blood Flow (Qa), when eEBF adjusts with Dynamic Arterial Line Pressure (DALP) in patients with Arteriovenous fistulae in hemodialysis treatment.

DETAILED DESCRIPTION:
Accesses that show a large (>15%) decrement over time in vascular access blood flow are associated with a high risk of thrombosis. Serial measurements of vascular access blood flow predict access thrombosis. At the moment, the measurement of access flow is time consuming, operator dependent, so that it cannot be done with every treatment. We hypothesized that extracorporeal blood flow at pressure of -200 to -260 mmHg in arterial line has correlation with access blood flow and this can be used to estimate access blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic Kidney Disease K-DIGO 5d in hemodialysis treatment)
* Permanent vascular accesses with native arteriovenous fistulas (AVF)
* AVF that were at least 12 weeks old

Exclusion Criteria:

* Inflammation and pain in AVF
* Negation to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic Kidney Dissease K-DIGO 5d in hemodialysis.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-03; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Acces Blood Flow | Acces Blood Flow
  Acces Blood Flow: cuantity of Blood that Flow throw venous acces in ml/min

CONTACTS AND LOCATIONS:
Overall Officials: Franklin B Mora, M.D., Principal Investigator — HOSPITAL JOSE CARRASCO ARTEAGA DEL INSTITUTO ECUATORIANO DE SEGURIDAD SOCIAL REGIONAL 3; Luis R Mariscal, M.D., Study Chair — Instituto Nacional de Cardiología Ignacio Chávez; Guadalupe C De la Cruz, R.N., Study Chair — Instituto Nacional de Cardiología Ignacio Chávez; Héctor G Pérez-Grovas, M.D., Study Chair — Instituto Nacional de Cardiología Ignacio Chávez; Fabián H Ortiz, MsC, Principal Investigator — Hospital Clínica Kennedy, Guayaquil Ecuador
Locations (1):
- Instituto Nacional De Cardiología Ignacio Chávez, Mexico City, Distrito Federeal, Mexico